CLINICAL TRIAL: NCT05464758
Title: The Effects of Cold Habituation on Peripheral Blood Flow, Hand Function, and Thermal Comfort
Brief Title: The Effects of Cold Adaptation on Skin Blood Flow, Hand Function, and Comfort in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-04H; MO210025 (Other Grant/Funding Number: USAMRDC Military Operational Medicine Research Program)
Record Dates: First submitted 2022-07-06; First posted 2022-07-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cold Exposure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cold habituation (Experimental): 8-day cold habituation
  Interventions: Other: Repeated cold exposure

INTERVENTIONS:
Other: Repeated cold exposure — 8 consecutive days of exposure to 8°C air for 120 minutes each day

SUMMARY:
In cold weather environments, blood flow to the extremities is significantly reduced, which severely impairs hand function and induces thermal discomfort. Prolonged or repeated cold exposure elicits an adaptive habituation response that is characterized by blunted skin vasoconstriction and thus may be an effective strategy to improve peripheral perfusion, reduce thermal discomfort, and maintain hand function during cold weather military operations. Since mission conditions often involve low ambient temperatures, countermeasures that reduce cold-induced decrements in hand function and thermal comfort are important to enhance Warfighter readiness in cold weather battlefield environments. The goals of this study are to 1) evaluate the effectiveness of cold habituation in improving skin blood flow, hand function, and thermal comfort during cold exposure and 2) identify the mechanisms that contribute to improvements in skin blood flow following habituation.

DETAILED DESCRIPTION:
Participants (n=15, 18-39 yrs) will complete a preliminary cold air exposure (baseline testing) followed by 8 days of repeated cold air exposures with minimal clothing. The cold exposures will be 2 hours in duration and will be conducted in 8°C (46°F) conditions. Before and after the repeated cold exposures, participants will undergo hand function tests, assessments of thermal comfort, and skin blood flow testing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-39
* In good health as determined by OMSO (Office of Medical Support and Oversight)
* Willing to refrain from exercise and caffeinated or alcoholic beverages for 12 hours before each testing session
* Willing to refrain from smoking or tobacco use 8 hours before each testing session

Exclusion Criteria:

* History of cold injuries of any severity (e.g., frostbite, trench foot, chilblains).
* Raynaud's syndrome.
* Cold-induced asthma/bronchospasm
* Previous hand/finger injuries that impair dexterity and hand function.
* Metal hardware (plates/screws) in the forearms and hands.
* Current use of medications or dietary supplements that could alter cardiovascular, thermoregulatory, or vascular control (e.g., anti-hypertensives, statins).
* Known allergies to medical adhesives.
* Heart, lung, kidney, muscle, or nerve disorder(s)
* A planned MRI during the study or within 2 days after completing a cold test.
* Women who are pregnant, planning to become pregnant, or breastfeeding.
* Not willing to have small areas of skin on the body shaved (if deemed necessary for attachment of study instrumentation)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Skin blood flow | 8 days
  Skin blood flow will be measured using non-invasive laser-Doppler flowmetry probes before and during cold exposure. Output (red blood cell flux) will be divided by mean arterial blood pressure to give an index of cutaneous vascular conductance [CVC, flux/mmHg].
Skin temperature | 8 days
  Skin temperatures [in °C] at up to 10 sites on the body will be measured using skin thermistors before and during cold exposure. Hand and foot skin temperatures will also be measured with a thermography imaging camera.
Manual dexterity - Pegboard | 3 days
  Pegboard scores will be obtained before and during cold exposure. Scores are the number of pegs placed into the boards.
Manual dexterity - Minnesota Rate of Manipulation | 3 days
  Minnesota Rate of Manipulation dexterity scores will be obtained before and during cold exposure. Scores are the time [in seconds] required to move small blocks various distances.
Hand and finger strength | 3 days
  Pinch and hand strength [in kg] will be measured using a pinch meter and grip strength device (dynamometer). Participants will complete three pinch strength tests and one grip strength test before and during cold exposure.
Cold perception | 5 days
  Ratings of thermal comfort, thermal sensation, and pain perception [in arbitrary units] will be assessed using visual analogue scales before and during cold exposure.

SECONDARY OUTCOMES:
Metabolic heat production | 5 days
  Oxygen consumption and carbon dioxide production [ml/kg/min] will be measured using computerized indirect calorimetry before and during cold exposure. Oxygen consumption and carbon dioxide production will be combined to report metabolic heat production in Watts per meter squared.
Body core temperature | 5 days
  Body core temperature [in °C] will be measured using a telemetry pill self-inserted as a suppository during cold exposure.
Blood pressure | 12 days
  Brachial artery blood pressure [in mmHg] will be measured using an automated blood pressure cuff before and during cold exposure.
Plasma norepinephrine | 3 days
  Circulating concentrations of norepinephrine [in pg/ml] will be assessed in blood collected via venipuncture before and after cold exposure.
Heart rate | 12 days
  Heart rate [in beats per min] will be measured using an automated cuff before and during cold exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Billie K Alba, Ph.D., Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- U.S. Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT05464758/ICF_000.pdf